CLINICAL TRIAL: NCT00046124
Title: Organophosphate Pesticides and Human Reproductive Health
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Other Study IDs: 8957-CP-001
Record Dates: First submitted 2002-09-20; First posted 2002-09-23 (Estimated); Last update posted 2006-09-04 (Estimated); Status verified 2006-09

CONDITIONS: Fecundability; Spermatazoa Disorders; Menstruation Disorders; Endocrine Dysfunction
MeSH Terms: conditions — Menstruation Disturbances

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
This prospective cohort study assesses the effects of exposure to organophosphate (OP) pesticides on adverse reproductive outcomes in both male and female agricultural workers in China. We will enroll women and their spouses, who are attempting to become pregnant, and observe reproductive endpoints including (1) semen parameters (concentration, total count, motility, progression and morphology), (2) menstrual disorders (oligomenorrhea, amenorrhea, polymenorrhea, intermenstrual bleeding, prolonged menstrual bleeding, dysmenorrhea, and irregular menstruation); (3) alterations in hormone patterns including reduced estrogen excretion (REE), anovulation, abnormal luteal phase (ALP), and abnormal follicular phase (AFP) in women and abnormalities of LH, FSH, TSH, SHBG, inhibin-B and testosterone in men; (4) fecundability; and (5) pregnancy outcomes including spontaneous abortion, preterm delivery, low birth weight, and intrauterine growth retardation.

ELIGIBILITY:
Inclusion Criteria:

* it must be the first marriage for both the woman and her husband and they must currently live in the study area;
* the female's age must range from 20 to 34 years;
* the couple has no plan to leave the study area in which they live for the next two years.

Exclusion Criteria:

* those who are currently pregnant;
* those who have tried unsuccessfully to get pregnant for at least 1 year;
* those who are current or former smokers;
* those who plan to move in the coming year.

Ages: 20 Years to 34 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Anhui Medical University, Anqing, Anhui, China